CLINICAL TRIAL: NCT00327847
Title: Optimizing Vitamin D Nutrition in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Winthrop University Hospital (Other)
Responsible Party: John F. Aloia, MD, Winthrop-University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB Protocol #04037
Record Dates: First submitted 2006-05-18; First posted 2006-05-19 (Estimated); Last update posted 2008-09-25 (Estimated); Status verified 2008-09

CONDITIONS: Vitamin D Deficiency
MeSH Terms: conditions — Vitamin D Deficiency

INTERVENTIONS:
Drug: Oral Vitamin D Supplementation

SUMMARY:
The purpose of this study is to determine the average dosage of oral vitamin D supplementation to maintain optimal vitamin D levels in the body and to see if there are differences in the response to oral vitamin D supplementation between African-American and Caucasian subjects.

DETAILED DESCRIPTION:
There is ample evidence that improvement in vitamin D nutrition retards bone loss and prevents fractures in the elderly. It is clear that many people living in areas of northern latitude have less than optimal levels of vitamin D. The current recommendations for vitamin D intake are not enough to bring a large majority of the population to the desired adequate level. Furthermore, differences have been observed in the amount of Vitamin D produced in the skin in whites and blacks.

Based on the evidence from literature and our experience from prior studies we hypothesize that:

1. the dose of oral vitamin D3 supplement exceeds current recommendations to achieve adequate desired level;
2. there may be differences in the dose-response to vitamin D supplement between Blacks and Whites; and
3. vitamin D supplementation that produces serum 25-hydroxyvitamin D (25-OHD) levels in the range proposed is safe.

The aims for this pilot study are to determine:

1. the average dose of vitamin D3 needed to attain 25-OHD levels between 80-140 nmol/L in a healthy population of mixed races; and
2. if there are differences in response to vitamin D3 supplementation between African American and Caucasians subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy African-American and Caucasian adults aged 18-65 years.

Exclusion Criteria:

* Subjects who are not either African-American or Caucasian. The investigators plan to examine racial differences in response to oral vitamin D dosing and, therefore, have chosen the most affected (African-American) and the least affected (Caucasian) racial groups. Including other racial/ethnic groups may confound the results unless they are studied as separate groups.
* Any chronic medical illness including diabetes mellitus, history of myocardial infarction or heart failure, malignancy, hypertension (systolic blood pressure [SBP] > 140), obesity (body mass index [BMI] > 35 kg/m2), history of anemia, leukemia, or other hematologic abnormalities, lupus, rheumatoid arthritis, or other rheumatologic disease, or kidney disease of any kind as determined by history and physical examination.
* Subjects with osteoporosis or taking medications for osteoporosis such as bisphosphonates.
* Pregnancy.
* Use of medication that influences bone metabolism (i.e. anticonvulsant medications, steroids, diuretics).
* Significant deviation from normal in either history, physical examination, or laboratory tests, as evaluated by the primary investigator.
* Patients with a history of hypercalciuria, hypercalcemia, nephrolithiasis, and active sarcoidosis.
* Participation in another investigational trial in the past 30 days prior to the screening evaluation.
* Unexplained weight loss of > 15% during the previous year or history of anorexia nervosa.
* Medications that interfere with vitamin D metabolism. Oral contraceptive use will be allowed, but will be appropriately documented.
* Smokers greater than 1 pack per day.
* Patients reporting alcohol intake greater than 2 drinks daily.
* Subjects with baseline 25-OHD level greater than 80 nmol/L or less than 20 nmol/L.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2004-12; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John F. Aloia, M.D., Principal Investigator — Winthrop University Hospital
Locations (1):
- Winthrop University Hospital, Mineola, New York, United States